CLINICAL TRIAL: NCT02316314
Title: Characterization of the Cardiac Phenotype of Friedreich's Ataxia (FRDA)
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1408015429
Record Dates: First submitted 2014-11-12; First posted 2014-12-12 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's Ataxia; Cardiomyopathy; FRDA; Ataxia
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies; Ataxia | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Amount: Up to 300 mL of blood will be collected for the entire study and up to 85 mL of blood will be collected for a single visit. (CBC = 5 mL per visit; Clotting = 6 mL per visit; Chemistry = 7 mL per visit; Liver function = 5 mL per visit; Cardiac enzymes = 5 mL per visit; Future serum = up to 20 mL per visit; Future plasma = up to 20ml per visit; Genetic analysis = 4 mL; HbA1c = 5mL; HIV test = 7 mL; and Anti-AAVrh.10 = 10 mL). An additional 10 ml of blood will be drawn after performing the CPET (5ml, 15 minutes +/- 15 minutes post CPET and another 5 ml 2 hours post CPET).
  Urine Amount: Approximately 36 mL of urine will be collected for the entire study and approximately 12 mL of urine will be collected for a single visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals diagnosed with FRDA: Individuals diagnosed with FRDA, to undergo the cardiac magnetic resonance imaging (CMR), exercise-stress test, echocardiogram (ECHO), and cardiac-related blood studies
  Interventions: Procedure: Cardiac magnetic resonance imaging (CMR); Procedure: Exercise-stress test; Procedure: Echocardiogram (ECHO); Procedure: Cardiac-related blood studies
- Healthy controls: Individuals without FRDA, to undergo the cardiac magnetic resonance imaging (CMR), exercise-stress test, echocardiogram (ECHO), and cardiac-related blood studies
  Interventions: Procedure: Cardiac magnetic resonance imaging (CMR); Procedure: Exercise-stress test; Procedure: Echocardiogram (ECHO); Procedure: Cardiac-related blood studies

INTERVENTIONS:
Procedure: Cardiac magnetic resonance imaging (CMR) — CMR is a non-invasive way to take a high-resolution image of the heart and vessels. CMR uses powerful magnets and radio waves to obtain the image. During the CMR, you will have a substance injected into your vein called "contrast" to get a better picture of the heart.
Procedure: Exercise-stress test — You will be asked to pedal on a bicycle with your arms to see how much work you can do and how far you can go.
Procedure: Echocardiogram (ECHO) — An echocardiogram is an ultrasound of the heart done at rest.
Procedure: Cardiac-related blood studies — The blood test involves drawing blood from a vein in the arm by placing a needle in it. The total amount of blood to be drawn for a single visit will be up to 57 mL (12 teaspoons).

SUMMARY:
Friedreich's ataxia (FRDA) is an autosomal recessive disease characterized by loss of coordination and cardiomyopathy. It is the most common form of inherited ataxia with an incidence in 1/50,000 in the Caucasian population. FRDA is associated with progressive damage to the nervous system, resulting in symptoms ranging from gait disturbance to speech problems, as well as diabetes and heart disease. The heart disease manifests as cardiomyopathy, and is responsible for approximately 60% of deaths from FRDA. This study is designed to characterize the cardiac manifestations of the disease using exercise, MRI, ECHO and serum parameters, in the context of the neurological disease. In addition, this study will demonstrate that corneal confocal microscopy (CCM) may also provide a biomarker for FRDA.

DETAILED DESCRIPTION:
The focus of this study is to assess cardiac dysfunction in individuals with FRDA using 4 modalities: hand crank exercise, cardiac magnetic resonance (CMR) imaging, echocardiography (ECHO), and serum measurements of cardiac status, including high sensitivity troponin, a measure of cardiac myocyte damage; N-terminal prohormone of brain natriuretic peptide (NTproBNP), a measure of heart failure; and creatine phosphokinase (CPK), a general measure of muscle damage. While there have been individual studies of some of these modalities, there are no studies that correlate these parameters and it is not known which parameters are more sensitive to cardiac dysfunction. This preliminary study will help define the parameters most useful in assessing the cardiac involvement in FRDA. In addition, the study will investigate noninvasive tests and procedures that may serve as biomarkers for the neurologic disease. In other neurological diseases, non-invasive examination of the number and structure of nerve cells in the cornea has been assessed as an indication of disease progression.

ELIGIBILITY:
Friedreich's Ataxia - Inclusion Criteria:

* Males and females, age 12 to 50
* Willing and able to provide informed consent (adolescents will need to provide assent and a parent to provide consent)
* Definitive diagnosis of FRDA, based on clinical phenotype and genotype
* Left ventricle ejection fraction measured by ECHO of >35% (If results of an ECHO are not available for a potential subject, then an ECHO will first be performed and subjects with an LVEF <35% will not be required to perform the CPET)

Friedreich's Ataxia - Exclusion Criteria:

* Signs and symptoms of cardiac failure
* Moderate to severe atrial or ventricular arrythmias
* History of angina pectoris
* Implanted pacemaker and/ or defibrillator or any other device that would preclude MRI assessment
* Any form of dialysis; Severe or end-stage CKD (CKD 4 or 5, eGFR < 30 ml/min/1.73 m2) without dialysis; eGFR 30 to 40 ml/min/1.73 m2 without dialysis; Acute kidney injury (If a recent assessment is not available, then a blood test to assess kidney function will be performed prior to cardiac MRI)
* Females who are pregnant
* Receipt of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to screening, or active enrollment in an investigational medication or device study
* Unable to undergo cardiac MRI with gadolinium contrast or claustrophobia
* Clinical history or evidence of Type 1 or Type 2 Diabetes mellitus
* Any condition, disorder, or abnormal laboratory test findings at screening which, in the judgment of the investigator, would interfere with the individual's ability to comply with all study requirements, or would require the administration of treatment during the study that could potentially affect the interpretation of the study data, or would place the individual at an unacceptable risk by his/ her participation in the study

Normal controls - Inclusion Criteria:

* Males and females, age 12 to 30
* Willing and able to provide informed consent (Adolescents will need to provide assent and a parent to provide consent)
* Matched age, gender and ethnicity to the FRDA group
* Capable of undergoing the various modalities of cardiac assessment
* Left ventricle ejection fraction measured by ECHO of >35% (If results of an ECHO are not available for a potential subject, then an ECHO will first be performed and subjects with an LVEF <35% will be withdrawn from the study)

Normal controls - Exclusion Criteria:

* Individuals not deemed in good overall health by the investigator will not be accepted into the study
* Signs and symptoms of cardiac failure
* Moderate to severe atrial or ventricular arrhythmias
* History of angina pectoris
* Implanted pacemaker and/ or defibrillator or any other device that would preclude MRI assessment
* Any form of dialysis; Severe or end-stage CKD (CKD 4 or 5, eGFR < 30 ml/min/1.73 m2) without dialysis; eGFR 30 to 40 ml/min/1.73 m2 without dialysis; Acute kidney injury (If a recent assessment is not available, then a blood test to assess kidney function will be performed prior to cardiac MRI)
* Females who are pregnant or lactating
* Receipt of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to screening, or active enrollment in an investigational medication or device study
* Unable to sit with back support
* Unable to undergo cardiac MRI with gadolinium contrast or claustrophobia
* Unable to undergo exercise tests
* Clinical history or evidence of Type 1 or Type 2 Diabetes mellitus
* Any condition, disorder, or abnormal laboratory test findings at screening which, in the judgment of the investigator, would interfere with the individual's ability to comply with all study requirements, or would require the administration of treatment during the study that could potentially affect the interpretation of the study data, or would place the individual at an unacceptable risk by his/ her participation in the study

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be composed of individuals with FRDA and individuals without FRDA. Individuals without FRDA will be age, gender and ethnicity matched to the individuals with FRDA.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Level of troponin, BNP, and CPK in blood | 30 minutes
  Average the levels of troponin for each subject
echocardiogram | 2 hour
  Evaluate the results of subject's Echo cardiograms
exercise-stress test | 2 hour
  Evaluate off the results of the exercise-stress test

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided